CLINICAL TRIAL: NCT01185379
Title: Investigation of the Effects of Efalex Active 50+ on Cognitive Performance, Well-being and Cerebral Hemodynamics in Healthy Adults Aged 50-70 Years Reporting Subjective Memory Deficits
Brief Title: The Effects of Efalex Active 50+ on Cognitive Performance, Well-being and Cerebral Hemodynamics in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Efamol Ltd (Industry)
Responsible Party: Principal Investigator, David Kennedy, Prof. David Kennedy, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 31N1
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2010-11

CONDITIONS: Cognitive Function; Mood; Well-being; Cerebral Blood Flow
Keywords: Docosahexaenoic acid; omega 3; cerebral blood flow; Near Infrared spectroscopy; cognitive function; mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Efalex Active 50+ (Active Comparator)
  Interventions: Dietary Supplement: Efalex active 50+
- DHA-rich fish oil (Active Comparator)
  Interventions: Dietary Supplement: DHA rich fish oil
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Efalex active 50+ — 4 x 500 mg Efalax Active 50+, to be taken daily for 6 months.
  Arms: Efalex Active 50+
Dietary Supplement: DHA rich fish oil — 4 x 500 mg DHA rich tuna oil to be taken daily for 6 months
  Arms: DHA-rich fish oil
Dietary Supplement: Placebo — 4 x 500 mg capsules to be taken daily for 6 months
  Arms: Placebo

SUMMARY:
Dietary intake of omega-3 polyunsaturated fatty acids (n-3 PUFAs) is inversely associated with cognitive decline and dementia (e.g. Kalmijn et al. 2004, Heude et al. 2003, Morris et al. 2005, Dullemeijer et al. 2009). Recently, the effects of supplemental docosahexaenoic acid (DHA) on behavioural outcomes in older adults has been explored, however two trials addressing this issue have published conflicting results regarding the efficacy of DHA supplementation, with one reporting a benefit of treatment on cognitive performance (Yurko-Mauro et al. 2010), while the other did not (Dangour et al. 2010).

One area of research that has yet to be explored in this cohort is the effects of n-3 PUFAs on brain function in physiological terms. It is also possible that n-3 PUFAs, in combination with other compounds, may be more beneficial than treatment with n-3 PUFAs in isolation. The current study will explore several separate hypotheses within the same cohort. These are that Efalex Active 50+ may have a beneficial effect on:

* Cognitive performance
* Mental fatigue in response to cognitively demanding tasks
* Self-reported mood/well-being
* Task-related cerebral blood flow response

The proposed study therefore has two aims; the primary aim is to evaluate the cognitive and mood/well-being effects of Efalex Active 50+, a dietary supplement containing a number of potentially cognition enhancing components including DHA, phosphatidylserine, vitamin B12, folic acid and Ginkgo biloba, compared with placebo in a sample of older adults aged 50-70 years (Cognitive Study). The second is to evaluate the cerebral haemodynamic effects of the same treatment formulation in a sample drawn from the same population, with the addition of a third DHA-only arm (Hemodynamics Study). The intervention period will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Aged 50-70 years
* Low consumer of oily fish (≤ 1 portion/month)
* Has not taken vitamin/herbal supplements in the past 3 months
* Has not taken omega-3 supplement (including cod liver oil) in the past 2 years
* Has a good level of written and spoken English
* Has an MMSE score > 24
* Is suffering from a memory complaint (MAC-Q score > 24)

Exclusion Criteria:

* BMI > 35
* Smokes more than 15 cigarettes per day
* History of alcohol/drug abuse
* Currently taking statins/antidepressant/blood thinning medication
* Has high blood pressure
* Suffers from migraines/anaemia/heart or lung disorder/diabetes/active infections/jaundice/haemophilia or other clotting disease
* Has learning difficulties/dyslexia/colour blindness
* Is HIV positive
* Has hepatitis

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 6 months
  Performance on a number of tasks assessing cognitive function across domains (attention, memory, executive function) will be measured.

SECONDARY OUTCOMES:
Cerebral Hemodynamics | 6 months
  Cerebral blood flow response to cognitive tasks will be assessed using Near Infrared Spectroscopy (NIRS). General cerebral blood flow will be assessed using Transcranial Doppler (TCD)
Mood/well-being | 6 months
  Mood and well-being will be assessed using a number of measures:
  Bond-Lader visual analogue scales, Profile of Mood States (POMS), General Health Questionnaire (GHQ), Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: David O Kennedy, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom